CLINICAL TRIAL: NCT07079761
Title: Facilitation of Extinction Retention and Reconsolidation Blockade by IV Allopregnanolone in PTSD.
Acronym: IV Allo PTSD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Ann M. Rasmusson, MD, Principal Investigar, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2025000693; 7R01MH122867-05 (NIH)
Record Dates: First submitted 2025-06-03; First posted 2025-07-23 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-07

CONDITIONS: Post Traumatic Stress Disorder
Keywords: Trauma; Allopregnanolone; Neurosteroid
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Wounds and Injuries | interventions — Pregnanolone; SBE7-beta-cyclodextrin; Sodium Chloride; SBE4-beta-cyclodextrin

STUDY DESIGN:
Intervention Model Description: Active drug vs. placebo will be administered in two separate experiments to a population of medically healthy, non-medicated patients with PTSD stratified by sex and by menstrual phase within female sex.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: In this double-blind, placebo controlled, randomized trial, active drug and matching placebo will be supplied by the research pharmacy. Participants, assessors, and the investigators will be blind to treatment condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- IV Allopregnanolone (Allo) for Extinction Retention (Expt. 1) (Experimental): Arm 1 of Expt. 1 includes women in the early follicular or mid-luteal phase of the menstrual cycle and men with PTSD who receive IV Allo immediately after completion of extinction training.
  Interventions: Behavioral: Experiment 1: Three-day aversive conditioning, extinction, and extinction retention testing paradigm; Drug: Allopregnanolone (Allo) with 6% USP Dexolve (sulfobutyl ether-beta-cyclodextrin sodium salt) in 0.9% saline for IV infusion will be provided by the University of California, Davis, GMP manufacturer.
- IV Placebo for Extinction Retention (Expt. 1) (Placebo Comparator): Arm 2 of Expt. 1 includes women in the early follicular or mid-luteal phase of the menstrual cycle and men with PTSD who receive IV placebo immediately after completion of extinction training.
  Interventions: Behavioral: Experiment 1. Three-day aversive conditioning, extinction, and extinction retention testing paradigm; Other: Matching IV Placebo
- IV Allo for Reconsolidation Blockade (Expt. 2) (Experimental): Arm 1 of Expt. 2 will include women in the early follicular or mid-luteal phase of the menstrual cycle and men with PTSD who receive IV Allo immediately after reactivation of the conditioned aversive memory by exposure to one conditioned stimulus (CS+).
  Interventions: Behavioral: Experiment 2. Three-day aversive conditioning, reconsolidation blockade, and testing paradigm; Drug: Allopregnanolone (Allo) with 6% USP Dexolve (sulfobutyl ether-beta-cyclodextrin sodium salt) in 0.9% saline for IV infusion will be provided by the University of California, Davis, GMP manufacturer.
- IV Placebo for Reconsolidation Blockade (Expt. 2) (Placebo Comparator): Arm 2 of Expt. 2 will include will include women in the early follicular or mid-luteal phase of the menstrual cycle and men with PTSD who receive IV placebo immediately after reactivation of the conditioned aversive memory by exposure to one conditioned stimulus (CS+).
  Interventions: Behavioral: Experiment 2. Three-day aversive conditioning, reconsolidation blockade, and testing paradigm; Other: Matching IV Placebo

INTERVENTIONS:
Behavioral: Experiment 1: Three-day aversive conditioning, extinction, and extinction retention testing paradigm — Day 1: Aversive conditioning will involve the pairing of a brief, noxious but not painful air blast to the neck (unconditioned stimulus; US) to a colored shape appearing on a computer monitor (conditioned stimulus). An auditory stimulus will serve as the startle probe. Day 2: Extinction training will occur followed by IV Allo administration. Day 3: The effects of IV Allo (administered on Day 2) on extinction retention as well as reinstatement of conditioned psychophysiological reactions will be assessed.
  Arms: IV Allopregnanolone (Allo) for Extinction Retention (Expt. 1)
Drug: Allopregnanolone (Allo) with 6% USP Dexolve (sulfobutyl ether-beta-cyclodextrin sodium salt) in 0.9% saline for IV infusion will be provided by the University of California, Davis, GMP manufacturer. — On Day 2 of Experiment 1, a 1.7 mcg/kg dose of IV Allo will be administered over 5 minutes at the completion of extinction training to raise resting plasma Allo plus pregnanolone (PA) levels by 1500 pg/ml. This will be followed by a 4-5-hour continuous infusion of IV Allo at 2.6 mcg/kg/hr to maintain resting plasma Allo levels at the target level.
  Other Names: U.S. P. equivalent: brexanolone (SAGE Therapeutics) (IV Allopregnanolone with Captisol)
  Arms: IV Allopregnanolone (Allo) for Extinction Retention (Expt. 1)
Behavioral: Experiment 1. Three-day aversive conditioning, extinction, and extinction retention testing paradigm — Day 1: Aversive conditioning will involve the pairing of a brief, noxious but not painful air blast to the neck (unconditioned stimulus; US) to a colored shape appearing on a computer monitor (conditioned stimulus). An auditory stimulus will serve as the startle probe. Day 2: Extinction training will occur followed by IV Allo administration. Day 3: The effects of IV Allo (administered on Day 2) on extinction retention as well as reinstatement of conditioned psychophysiological reactions will be assessed.
  Arms: IV Placebo for Extinction Retention (Expt. 1)
Other: Matching IV Placebo — On Day 2 of Experiment 1, participants randomized to placebo will receive IV matching placebo over 5 minutes at the completion of extinction training followed by a continuous infusion of matching placebo over the next 4-5 hours. The matching IV placebo will be administered according to the same per kg dosing regimen as that for active drug.
  Other Names: 6% USP Dexolve alone in 0.9% saline for IV infusion will be provided by the University of California, Davis, GMP manufacturer.
  Arms: IV Placebo for Extinction Retention (Expt. 1)
Behavioral: Experiment 2. Three-day aversive conditioning, reconsolidation blockade, and testing paradigm — Day 1: Aversive conditioning will involve the pairing of a brief, noxious but not painful air blast to the neck (unconditioned stimulus; US) to a colored shape appearing on a computer monitor (conditioned stimulus). An auditory stimulus will serve as the startle probe. Day 2: Brief exposure to the conditioned stimulus will be followed by IV Allo administration. Day 3: The effects of IV Allo (administered on Day 2) on reconsolidation blockade and reinstatement of conditioned psychophysiological reactions will be assessed.
  Arms: IV Allo for Reconsolidation Blockade (Expt. 2)
Drug: Allopregnanolone (Allo) with 6% USP Dexolve (sulfobutyl ether-beta-cyclodextrin sodium salt) in 0.9% saline for IV infusion will be provided by the University of California, Davis, GMP manufacturer. — On Day 2 of Experiment 2, a 28 mcg/kg dose of IV Allo will be infused over 30 minutes following brief reactivation of aversively conditioned psychophysiological reactions, after which IV fluid only (0.9% normal saline) will be administered over 4-5 hours.
  Other Names: U.S. P. equivalent: brexanolone (SAGE Therapeutics) (IV Allopregnanolone with Captisol)
  Arms: IV Allo for Reconsolidation Blockade (Expt. 2)
Behavioral: Experiment 2. Three-day aversive conditioning, reconsolidation blockade, and testing paradigm — Day 1: Aversive conditioning will involve the pairing of a brief, noxious but not painful air blast to the neck (unconditioned stimulus; US) to a colored shape appearing on a computer monitor (conditioned stimulus). An auditory stimulus will serve as the startle probe. Day 2: Brief exposure to the conditioned stimulus will be followed by IV Allo administration. Day 3: The effects of IV Allo (administered on Day 2) on reconsolidation blockade and reinstatement of conditioned psychophysiological reactions will be assessed.
  Arms: IV Placebo for Reconsolidation Blockade (Expt. 2)
Other: Matching IV Placebo — On Day 2 of Experiment 2, matching IV placebo will be infused over 30 minutes following brief reactivation of aversively conditioned psychophysiological reactions, after which IV fluid only (0.9% normal saline) will be administered over the 4-5 hours. The matching IV placebo will be administered according to the same per kg dosing regimen as that for active drug.
  Other Names: 6% USP Dexolve alone in 0.9% saline for IV infusion will be provided by the University of California, Davis, GMP manufacturer.
  Arms: IV Placebo for Reconsolidation Blockade (Expt. 2)

SUMMARY:
Purpose: About 6.4% of the U.S. population suffers from posttraumatic stress disorder (PTSD). Trauma-focused psychotherapies are generally effective in PTSD, but responses vary greatly across individuals and PTSD subpopulations. Neurobiological factors impacted by life experiences, stress, and genetics can affect treatment responses. These factors can alter brain capacities needed to reprocess traumatic memories prevent them from triggering intensely distressing, disruptive, out-of-place responses.

For example, during psychotherapy for PTSD, trauma memory activation engages two competing brain processes that affect recovery: "extinction" versus "reconsolidation" of trauma-related emotional, physiological, and behavioral responses. This study tests whether a single intravenous (IV) dose of allopregnanolone (Allo) compared to placebo (which is non-active): promotes consolidation of extinction learning (sub-study 1) or blocks reconsolidation of physiological responses triggered by aversive memories (sub-study 2). The study also tests whether Allo compared to placebo affects retention of non-aversive memories.

DETAILED DESCRIPTION:
Background: Allo is a neurosteroid (hormone) produced from progesterone by the brain, adrenal glands, testes, and ovaries. Production of Allo and its equally potent, structurally similar stereoisomer pregnanolone (PA) is stimulated when certain neurons in the brain are activated and when stress activates the adrenal glands. Allo and PA markedly increase effects of gamma-amino-butyric acid (GABA; an inhibitory neurotransmitter) in the brain, thereby regulating arousal and responses to stress. Allo and PA also influence processes that strengthen or weaken memories.

Basic research suggests that several factors can reduce production of Allo: exposure to chronic or extreme stress, prolonged social isolation, chronic intermittent heavy alcohol use, certain oral contraceptives, chronic use of some psychiatric medications or other substances used to manage PTSD such as nicotine, exposure to environment toxins, and genetic predisposition.

Research shows that Allo and PA production is reduced in a large subpopulation of women and men with PTSD. Reduced Allo and PA is strongly associated with PTSD severity and poor retention of extinction learning, both of which contribute to chronic PTSD. The proposed study thus will be conducted in adult men and women with chronic PTSD. Women will be studied during two distinct phases of the menstrual cycle because progesterone levels (and therefore levels of Allo and PA) change markedly across the menstrual cycle, as do problems with extinction retention.

Study Procedures: Eligible participants between 18 and 55 years of age will take part in a widely used, standardized 3-day laboratory psychophysiology paradigm during which activation of the sympathetic nervous system (fight/flight system) is monitored via small electrode patches placed on the skin. The paradigm involves startle testing on Days 1, 2 and 3. During startle testing, participants will hear sudden bursts of white noise through headphones, see colored shapes on a computer screen, and feel sudden (not painful) blasts of air to the neck. The electrodes record participants' eye blinks, skin conductance, and heart rate. The startling sounds will be about as loud as a train but last only a fraction of a second. Participants will sit quietly with their eyes open as they listen. On study Day 2, participants are randomized by "luck of the draw" or "chance" to receive either IV Allo or placebo. On study Days 2 and 3, a brief memory test also will be conducted. Blood is collected each day for measurement of Allo, PA and other neurobiological factors that may affect the potential beneficial effects of Allo. There will be a follow up phone session (about a week after the Day 3 visit/session).

Before starting the above studies, the investigators will conduct pharmacokinetic (PK) studies in a small group of individuals with PTSD to confirm that the selected IV Allo doses increase blood Allo levels as expected.

Implications: These studies may help us understand treatable factors that increase risk for chronic or treatment-resistant PTSD and PTSD-related depression. They may also tell us whether treatments that increase Allo might help prevent or treat PTSD. IV Allo (brexanolone) at much higher doses than used in this study) is currently FDA-approved for the treatment of postpartum depression, supporting the potential for this research to spur development of Allo as a new treatment for PTSD.

Study Population: About 96 individuals with PTSD (between 18-55 years of age) will be recruited to participate in these studies. Half of the women will be studied during the follicular phase of the menstrual cycle (after onset of menses) and half during the luteal phase (after ovulation). The study is being conducted at Massachusetts General Hospital, Boston, MA.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 55 (at time of enrollment), reproductively mature, and English speaking.
* Meet criteria for chronic PTSD (i.e., CAPS-5 determined PTSD duration more than 3 months).
* Generally healthy and not on any prohibited medications (that could affect study outcomes).
* Willing to abstain from alcohol for 2 weeks and from nicotine, marijuana or illicit drugs for 4 weeks before experimental procedures and throughout the study.
* For biological females:

  * Natural menstrual cycle.
  * If of childbearing potential, female and partner must use 2 types of effective birth control (except for hormonal contraceptives, unless IUD or a device like Nuvaring) for a week before the IV Allo or placebo infusion, and for one month after.

Exclusion Criteria:

* Present an imminent risk to self or others or require clinical intervention to maintain safety
* Diagnosis of moderate or severe substance use disorder within three months of screening per administration of the DIAMOND substance abuse evaluation. Diagnosis of a mild substance use disorder within three months of screening will be allowed if the participant agrees to abstain from illicit drugs for one month and/or alcohol for 2 weeks prior to the experimental procedures, has a negative screening or follow-up urine toxicology and/or saliva alcohol test (if the screening test is positive), and tests negative for these substances on the morning of the experimental procedures.
* Bipolar I disorder, schizophreniform disorders, or clinically significant psychotic symptoms apart from the presence of trauma-related sensory hallucinations or negative beliefs.
* History of a suicide attempt within 1 year of enrolling.
* A history of severe TBI is exclusionary for the PK-1 and PK-2 studies. A history of moderate or severe TBI is exclusionary for the main studies (i.e., Expt. 1 and Expt. 2).
* Diagnosis of sleep apnea
* Awake resting O2 saturation < 96%
* Severe renal failure with an eGFR <30 ml/min
* Use of medications or substances (by report or toxicology testing) will be exclusionary under the following conditions:

  1. During screening for eligibility:

     1. Use of illicit substances, as well as prescribed opiates or benzodiazepines (either reported or detected on urine toxicology testing) will be exclusionary.
     2. Reported non-dependent use of cannabinoids or nicotine (indicated by a positive urine toxicology or cotinine test at screening) will not be exclusionary if the individual agrees to abstain from cannabinoids and nicotine for one month prior to the experimental procedures, has a follow-up negative screening test, and tests negative for these substances on the mornings of experimental procedures.
     3. A positive urine alcohol test at medical screening (which indicates uncontrolled alcohol use and likely moderate to severe alcohol dependence) will be exclusionary.
     4. A high serum gamma-glutamyl-transferase (GGT) test at screening (indicative of more remote recent drinking but not necessarily moderate to severe alcohol use or dependence) will not be exclusionary if the individual does not meet criteria for a moderate or severe alcohol use disorder within three months of screening, agrees to abstain from drinking for 2 weeks prior to the experimental procedures, and has normal follow-up urine alcohol and serum GGT tests.
     5. Use of non-illicit over the counter or prescribed medications that may increase the risk of IV Allo side effects or adversely affect the experimental results is exclusionary. Participants may agree to stop non-psychotropic medications used on a prn basis, such as acetaminophen, ibuprofen, or loratadine (a CYP3A inhibitor) for 5 half-lives of the parent drug or active metabolite (whichever is longer) before the experimental procedures. Regular psychotropic medications (including those used to treat non-psychiatric conditions, such as alpha1-antagonists prescribed for hypertension or urinary hesitancy) may be discontinued under the management of the potential participant's non-study prescriber for 3 months before evaluation for eligibility and participation in subsequent experimental procedures.
  2. On the mornings of the PK-1, PK-2, Expt. 1 or Expt. 2 experimental procedures:

     1. Use of any medications or substances that may increase the risk of IV Allo side effects or adversely affect the experimental results (indicated by report, urine toxicology, urine nicotine/cotinine testing, or urine alcohol testing) will be exclusionary.
     2. Systemic hormone therapy or contraception will be exclusionary [Exception: Hormonal IUDs (e.g., Mirena, Kyleena, Liletta, and Skyla) or other contraceptive devices (e.g., Nuvaring)] will be allowed if the participant still has normal menstrual periods and is found to ovulate using commercial urine test kits provided by study).
* Pregnancy (urine pregnancy tests given at each in-person session).
* Breast-feeding.
* Unable to tolerate IV placement or blood drawing by needle stick.
* Wear hearing aid(s) (For Expt. 1 and 2, not PK studies).
* Fail hearing test (For Expt. 1 and 2, not PK studies).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-08-04 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Experiment 1: Extinction retention | Day 3
  Extinction retention is calculated as a) the difference between the average skin conductance response (SCR) to the first 4 aversively conditioned stimulus (CS+) trials and the average SCR to first 4 neutral conditioned stimulus (CS-) trials on Day 3 minus b) the difference between the average SCR to the last 4 CS+ trials and last 4 CS- trials on Day 2.
Experiment 2: Reconsolidation blockade | Day 3
  Reconsolidation blockade will be assessed by calculating the average fear potentiated startle (FPS) response to the first 4 CS+ trials on Day 3. Lower scores indicate better reconsolidation blockade.

SECONDARY OUTCOMES:
Experiment 1: Reinstatement of conditioned fear | Day 3
  Reinstatement of conditioned fear will be assessed by calculating the average SCR to the last 4 CS+ trials minus the average SCR to the last 4 CS- trials on Day 3.
Experiment 2: Reinstatement of conditioned fear | Day 3
  Reinstatement of conditioned fear will be assessed as the average FPS to the last 4 CS+ trials on Day 3. Higher scores indicate greater reinstatement of conditioned fear.
Reinstatement of Conditioned Fear in Expt. 1 | Day 3
  Reinstatement of conditioned fear will be defined as the average SCR to the last 4 CS+ trials minus the average SCR to the last 4 CS- trials. For FPS, the last 4 CS+ trials will be examined. Higher scores indicate greater reinstatement of conditioned fear.
Reinstatement of Conditioned Fear in Expt. 2 | Day 3
  Reinstatement of conditioned fear will be defined as the average SCR to the last 4 CS+ trials minus the average SCR to the last 4 CS- trials. For FPS, the last 4 CS+ trials will be examined. Higher scores indicate greater reinstatement of conditioned fear.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States